CLINICAL TRIAL: NCT02647541
Title: Preoperative Nutritional Intervention and Outcomes Postoperative of Children Submitted to Heart Surgery for Congenital Heart Diseases
Brief Title: Preoperative Nutritional Intervention and Outcomes of Children Submitted to Heart Surgery for Congenital Heart Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thatiane Danielly Santos, RD, MSc, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TSantos
Record Dates: First submitted 2015-12-10; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Congenital Heart Disease; Malnutrition
Keywords: Children; Congenital heart disease; Nutritional status; Bioelectrical impedance
MeSH Terms: conditions — Heart Defects, Congenital; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional intervention (Experimental): Consultation with a dietitian, including nutritional recommendations and supplementation.
  Interventions: Dietary Supplement: Nutritional intervention
- Standard therapy (No Intervention): No specific nutritional recommendations.

INTERVENTIONS:
Dietary Supplement: Nutritional intervention — Consultation with a dietitian, nutritional recommendations to achieve the expected energy expenditure, with or without supplementation with enriched formulas.
  Arms: Nutritional intervention

SUMMARY:
The hypothesis of this study is a nutrition preoperatively in infants and children undergoing elective cardiac surgery with cardiopulmonary bypass leads to improvement in nutritional status, intervention, and that this results in good postoperative results.

DETAILED DESCRIPTION:
If this hypothesis is confirmed, there will be subsidies for systematic implementation of nutritional interventions in patients seen in service.

ELIGIBILITY:
Inclusion Criteria:

* Patient with congenital heart disease requiring elective surgical correction;
* Age> 30 days and ≤ 5 years, with the aim of excluding the neonatal period, which are operated children with complex heart defects, and older children, where the time living with the disease damages the myocardium and the pulmonary circulation, leaving only children with fewer serious and, in general, are less subjected to complex surgery diseases.

Exclusion Criteria:

* Chronic gastrointestinal diseases (defects, malabsorption, celiac disease, inflammatory bowel disease, diabetes mellitus);
* Patients with other organic defects that may compromise the growth and / or nutritional status;
* Patients undergoing emergency surgery;
* Request of parents or guardians at any time;
* Patients receiving exclusive breastfeeding;
* Died during the study period;
* Patients using cardiac pacemaker or other electrical or electronic device that interferes with the reading of the electrical bioimpedance.

Ages: 30 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 30 to 45 days prior to surgery
  Weight-for-age z-score

SECONDARY OUTCOMES:
Surgical outcomes | on average 15 days after surgery
  Length-of-hospital-stay

CONTACTS AND LOCATIONS:
Overall Officials: Thatiane D Santos, Msc, Principal Investigator — FMRP/USP
Locations (1):
- Faculty of Medicine of Ribeirão Preto / USP, Ribeirão Preto, São Paulo, Brazil